CLINICAL TRIAL: NCT00371761
Title: An Open-Label, Randomized, Comparative Study With PegIntron vs. Adefovir in the Treatment of Chronic Hepatitis B (CHB) e Antigen Positive Patients in Taiwan
Brief Title: PegIntron Versus Adefovir in the Treatment of Chronic Hepatitis B (CHB) e Antigen Positive Patients in Taiwan (P04498/MK-4031-278)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04498
Record Dates: First submitted 2006-08-31; First posted 2006-09-04 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis B, Chronic (CHB)
Keywords: Hepatitis B virus; Pegylated interferon alfa-2b (PegIntron)
MeSH Terms: conditions — Hepatitis B; Bronchiolitis Obliterans Syndrome | interventions — peginterferon alfa-2b; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PegIntron (Experimental): PegIntron, 1.5 micrograms/kg weekly, for up to 24 weeks followed by a 48-week observation phase
  Interventions: Biological: Pegylated interferon alfa-2b (PegIntron)
- Adefovir (Active Comparator): Adefovir, 10 mg daily, for up to 48 weeks followed by a 24-week observation phase
  Interventions: Drug: Adefovir dipivoxil (adefovir)

INTERVENTIONS:
Biological: Pegylated interferon alfa-2b (PegIntron) — Powder for injection in vials ( 100, and 120 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for up to 24 weeks
  Other Names: SCH 54031, Peg-Intron
  Arms: PegIntron
Drug: Adefovir dipivoxil (adefovir) — 10 mg adefovir dipivoxil (equivalent to 5.4.5 mg adefovir) tablets, oral, dose of 1 tablet per day for up to 48 weeks
  Other Names: Hepsera
  Arms: Adefovir

SUMMARY:
This is an open label, randomized, comparative, multi-center study. Subjects will be screened within 2 weeks prior to study entry to establish eligibility. Subjects who meet all the selection criteria will be randomly assigned 1:1 to (1) once-a-week, subcutaneous Pegylated interferon alfa-2b (PegIntron) (1.5 mcg/kg body weight) or (2) oral adefovir 10 mg daily. The treatment phase will be 24 weeks for PegIntron and 48 weeks for adefovir. All subjects completing the assigned treatment phase will be followed up for an additional 48 weeks for PegIntron and 24 weeks for adefovir as observation phase. The primary objective is to establish the efficacy profile of PegIntron. Secondary objectives are to compare the efficacy profile of PegIntron with that of adefovir, compare efficacy of PegIntron in lamivudine-naïve and lamivudine-experienced subjects, and to establish the safety profile of PegIntron in treating patients with hepatitis B e antigen (HBeAg)-positive chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, 18 to 70 years of age.
* Documented positive serum hepatitis B surface antigen (HBsAg) for a minimum of 6 months prior to randomization.
* Hepatitis B virus (HBV) replication and hepatitis documented by:

  * Serum HBV DNA (Hepatitis B Virus Deoxyribonucleic acid) >= 10^5 copies/mL within 3 months prior to entry
  * Positive serum hepatitis B e antigen (HBeAg) within 3 months prior to entry
  * Documented presence of ALT (Alanine Aminotransferase) twice (1 month apart) within 3 months prior to entry (2 to 10 folds above the upper normal level)
  * Liver biopsy finding shows evidence of chronic hepatitis without liver cirrhosis, document acceptable if no anti-HBV treatment within 1 year prior to randomization
  * Naïve or exposed to lamivudine (3 months treatment-free interval prior to randomization)
  * Adequate renal function (creatinine within normal upper limit).
* Compensated liver disease with certain minimum hematological and serum biochemical criteria.
* Thyroid stimulating hormone (TSH) and free T4 within normal ranges.
* Negative antibody to hepatitis C and hepatitis D.
* Negative antibody to human immunodeficiency virus.
* Negative evidence for hepatocellular carcinoma by alfa-fetoprotein and ultrasound within 1 month prior to randomization.

Exclusion Criteria:

* Women who are pregnant or nursing.
* Prior treatment for hepatitis with any interferon or adefovir, or other investigational anti-virus agents.
* Prior treatment for hepatitis with immunomodulatory drug within 2 years prior to randomization.
* Suspected hypersensitivity to interferon or adefovir.
* Liver cirrhosis.
* History of severe psychiatric disease, especially depression.
* Concurrent malignancies (including hepatocellular carcinoma).
* Unstable or significant cardiovascular diseases.
* Prolonged exposure to known hepatotoxins.
* History of thyroid disease poorly controlled on prescribed medication.
* Poorly controlled diabetes mellitus.
* Have suspected or confirmed significant hepatic disease from an etiology other than HBV.
* Severe renal disease or myeloid dysfunction.
* History of organ transplantation other than cornea and hair transplant.
* Any medical condition requiring chronic systemic administration of steroids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PegIntron | Adefovir
Started | 13 | 12
Completed | 5 | 2
Not Completed | 8 | 10
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Investigator Judgment | 2 | 3
Not completed — Study termination | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PegIntron | Adefovir | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.5) | 36.7 (13.6) | 36.7 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  Taiwan, Province Of China | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Combined Response Consisting of All Three Responses - (a) Serological Response, (b) Virological Response, and (c) Biochemical Response
Description: 1. Serological response is defined as Loss of HBeAg (Hepatitis B e antigen) and Appearance of anti-HBe (Hepatitis B e antibodies); participant is HBeAg negative and anti-HBe positive.
  2. Virological response was defined as having < 10^5 copies/mL of serum HBV DNA (Hepatitis B Virus Deoxyribonucleic Acid) by real-time PCR (Polymerase Chain Reaction).
  3. Biochemical response was defined as acheiving normal levels of ALT (Alanine Aminotransferase) level in Units/L.
Time Frame: At Week 72 [for Pegylated interferon alfa-2b (PegIntron), at 48 weeks post PegIntron treatment for up to 24 weeks; for Adefovir, at 24 weeks post adefovir treatment for up to 48 weeks]
Measure: Number; unit: Participants
Arm/Group | PegIntron | Adefovir
Number analyzed (Participants) | 13 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | PegIntron | Adefovir
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/12
Other Adverse Events (participants affected / at risk) | 13/13 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron (N=13) | Adefovir (N=12)
LAPAROSCOPIC SURGERY (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron (N=13) | Adefovir (N=12)
LEUKOPENIA (Blood and lymphatic system disorders) | 5 (9) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (2) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 4 (4) | 1 (1)
REGURGITATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 2 (3) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (2)
CHILLS (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 2 (2) | 0 (0)
FEELING COLD (General disorders) | 2 (3) | 0 (0)
FEELING HOT (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 1 (12) | 0 (0)
PYREXIA (General disorders) | 9 (63) | 0 (0)
FOOD ALLERGY (Immune system disorders) | 0 (0) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 2 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (6) | 1 (2)
ALPHA 1 FOETOPROTEIN INCREASED (Investigations) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (4) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (4) | 0 (0)
HAEMOGLOBIN INCREASED (Investigations) | 0 (0) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1)
VITAMIN C INCREASED (Investigations) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
ANOREXIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
FASCIITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
HAEMANGIOMA OF LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
HEADACHE (Nervous system disorders) | 4 (26) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DENTAL CARE (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator and Institution agree not to publish or publicly present any interim results of the study. Principal Investigator and Institution further agree to provide 45 days written notice to Sponsor prior to submission for publication or presentation to permit Sponsor to review drafts of abstracts and manuscripts for publication.